CLINICAL TRIAL: NCT03687502
Title: The Role of Contrast Enhanced Ultrasound in The Diagnosis of Children With Appendicitis
Brief Title: The Role of Contrast Enhanced Ultrasound in Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Tolulope Oyetunji, MD, Director, Health Outcomes Research, Department of Surgery, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Study00000329
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Masking Description: The CEUS image will be read at a future time by a Children's Mercy Hospital radiologist blinded to the results of the gray scale ultrasound and computed tomography (CT) scan if one was obtained; these will be used for comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): IV sulfur hexafluoride lipid-type A microspheres, 0.03 mL/kg, up to 2 doses per examination, total dose not to exceed 4.8 mL. Single examination per patient.
  Interventions: Drug: Sulfur hexafluoride lipid-type A microspheres

INTERVENTIONS:
Drug: Sulfur hexafluoride lipid-type A microspheres — Contrast Enhanced Ultrasound of the appendix
  Other Names: Lumason

SUMMARY:
This study seeks to determine the efficacy of Contrast Enhanced Ultrasound (CEUS) in improving the diagnosis of acute appendicitis in children, when compared to the standard grey-scale ultrasound.

DETAILED DESCRIPTION:
This will be a single-center, non-randomized trial that will add to our institution's current diagnostic algorithm using Contrast Enhanced Ultra Sound (CEUS) in subjects who are clinically suspicious for acute appendicitis.

For those who consent to study participation, we propose obtaining a CEUS after the initial gray-scale ultrasound. Once the initial ultrasound is complete, the contrast Lumason® (sulfur hexafluoride lipid type-A microspheres) will be administered through an already existing IV catheter and an abdominal scan will be completed. The patient will then continue with standard of care treatment per his treating physician. The CEUS image will be read at a future time by a Children's Mercy Hospital radiologist blinded to the results of the gray scale ultrasound and computed tomography (CT) scan if one was obtained; these will be used for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Present to Children's Mercy Adele Hall campus with a clinical concern for acute appendicitis
* Age 8 through 17 years
* seen between Institutional Review Board (IRB) approval date and 12/31/2019
* Seen Monday- Friday between the hours of 9:00 a.m. and 4:00 pm
* Has had an IV catheter placed as part of their standard of care

Exclusion Criteria:

* Known cardiac abnormality
* Pulmonary hypertension
* Known sensitivity to sulfur hexafluoride, polyethylene glycol 4000, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na), or palmitic acid
* Does not had an IV catheter placed
* Unable to roll over
* Unable to assent
* Pregnant
* Lactating
* Received an ultrasound image from a referring facility

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tolulope Oyetunji, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 37
Completed | 35
Not Completed | 2
Not completed — IV was removed prior to radiology visit for ultrasound | 1
Not completed — Lumason not available | 1

BASELINE CHARACTERISTICS:
Population: Subjects who completed both the greyscale and contrast enhanced ultrasound.
Groups:
- Contrast Enhanced Ultrasound Group: IV sulfur hexafluoride lipid-type A microspheres, 0.03 mL/kg, up to 2 doses per examination, total dose not to exceed 4.8 mL. Single examination per patient.
  Sulfur hexafluoride lipid-type A microspheres: Contrast Enhanced Ultrasound of the appendix
Arm/Group | Contrast Enhanced Ultrasound Group
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.4 [10 to 14.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26
  Black | 2
  Hispanic | 3
  Multiracial | 3
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Children With an Accurate Diagnosis of Appendicitis.
Description: Number of children with an accurate diagnosis of appendicitis when compared to the standard grey scale ultrasound and/ or CT scan based on the following categories:
  Category 1: Normal appendix Category 2: Appendix not fully visualized without secondary signs Category 3: Appendix not fully visualized with secondary signs Category 4: Appendicitis
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast Enhanced Ultrasound Group
Number analyzed (Participants) | 35
Participants
  Category 1 | 6
  Category 2 | 15
  Category 3 | 1
  Category 4 | 13

2. Secondary Outcome: Definitive Diagnosis
Description: Proportion of children with definitive diagnosis of appendicitis with use of CEUS.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast Enhanced Ultrasound Group
Number analyzed (Participants) | 35
Participants | 13

3. Secondary Outcome: Number of Participants Who Required Additional CT Scan
Description: "Number of Participants who Required Additional CT Scan"
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 35
Participants | 0

4. Secondary Outcome: Percentage of Negative Appendectomies
Description: Percentage of negative appendectomies
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast Enhanced Ultrasound Group
Number analyzed (Participants) | 35
Participants | 1

5. Secondary Outcome: Total Cost Difference Compared to Traditional Ultrasound
Description: Costs in comparison to traditional ultrasound
Time Frame: 60 days
Measure: Number; unit: Dollars
Arm/Group | Contrast Enhanced Ultrasound Group
Number analyzed (Participants) | 35
Dollars | 16

6. Secondary Outcome: Total Cost Difference Between Traditional Ultrasound in Comparison to Costs in CT Scan.
Description: Comparing total costs difference between traditional ultrasound in comparison to costs in CT scan.
  Total CT Scan Costs - Total Ultrasound Costs = Cost Difference.
Time Frame: 60 days
Measure: Number; unit: Dollars
Arm/Group | Contrast Enhanced Ultrasound Group
Number analyzed (Participants) | 35
Dollars | 6198

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03687502/Prot_000.pdf